CLINICAL TRIAL: NCT04452695
Title: Acceptability of Telehealth Triage Using Robotic Systems in COVID-19
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Peter R Chai, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2020P000957
Record Dates: First submitted 2020-06-29; First posted 2020-06-30 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: COVID-19; Telemedicine; Robotics; Emergencies; Emerging Infectious Disease
MeSH Terms: conditions — COVID-19; Emergencies; Communicable Diseases, Emerging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention arm: Patients presenting to the emergency department are triaged using a novel robotic telehealth triage system. Once triage is complete, patients complete a quantitative assessment to measure their acceptance and willingness to interact with the robotic telehealth system.
  Interventions: Device: Doctor Spot

INTERVENTIONS:
Device: Doctor Spot — Robotic platform (Boston Dynamics) controlled by clinician with video interface to facilitate telemedicine triage

SUMMARY:
The overall objective of this investigation is to understand the patient response to a robotic platform used to facilitate telehealth triage in the emergency department during the COVID-19 pandemic. The COVID-19 pandemic has altered the manner in which emergency department triage is completed. Attempts at cohorting individuals with potential COVID-19 disease in order to prevent disease transmission to healthcare workers and minimize the use of personal protective equipment (PPE) have renewed interest in telemedical solutions as a method to triage and manage individuals with COVID-19. This investigation deploys a legged robotic platform to facilitate agile, highly mobile telemedicine to manage COVID-19 patients in the emergency department. The primary objective is to measure the patient response to interacting with these systems.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the emergency department for evaluation
* > 18 years old

Exclusion Criteria:

* Brought to emergency department via ambulance
* <18 years old
* non-english speaking
* in extremis, or unable to participate due to underlying acute medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Acceptance of robotic telehealth system | Immediately after completion of triage
  Quantitative questionnaire on the acceptance of virtual robotic care graded on a likert scale (higher scores better)
Willingness to interact with robotic telehealth system | Immediately after completion of triage
  Quantitative questionnaire on the willingness to use this system again based on a likert scale (higher scores better)
Satisfaction of interacting with a robotic telehealth system | Immediately after completion of triage
  Quantitative questionnaire on the user satisfaction with their triage experience (How satisfied were you with your experience interacting with the robotic system today?)

SECONDARY OUTCOMES:
Use of robotic system versus in-person triage | Immediately after completion of triage
  Quantitative questionnaire comparing robotic triage process with in-person triage: Do you think your interaction with the robotic system was better, the same or no different than an in-person evaluation?)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chai PR, Dadabhoy FZ, Huang HW, Chu JN, Feng A, Le HM, Collins J, da Silva M, Raibert M, Hur C, Boyer EW, Traverso G. Assessment of the Acceptability and Feasibility of Using Mobile Robotic Systems for Patient Evaluation. JAMA Netw Open. 2021 Mar 1;4(3):e210667. doi: 10.1001/jamanetworkopen.2021.0667. PMID 33662134
- [Result] Huang HW, Chen J, Chai PR, Ehmke C, Rupp P, Dadabhoy FZ, Feng A, Li C, Thomas AJ, da Silva M, Boyer EW, Traverso G. Mobile Robotic Platform for Contactless Vital Sign Monitoring. Cyborg Bionic Syst. 2022;2022:9780497. doi: 10.34133/2022/9780497. Epub 2022 Apr 30. PMID 35571871